CLINICAL TRIAL: NCT05708716
Title: A Multi-component Non-pharmacological Intervention to Improve Cognitive Outcomes in Hematologic Cancer Survivors
Brief Title: Diet and Cognitive Training in Hematologic Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Noha Mohamed Sharafeldin, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 161221006; R03CA270671 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-02-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Impairment; Hematologic Malignancy
Keywords: Hematologic Cancer Survivors; Blood or Marrow Transplantation; Cognitive Training; Modified Ketogenic Diet
MeSH Terms: conditions — Cognitive Dysfunction; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet and Cognitive Training (Experimental): The arm will follow a modified ketogenic diet using an exogenous ketogenic formula (KetoCal) and use the online cognitive training program Lumosity at time of enrollment on the study.
  Interventions: Behavioral: Modified ketogenic diet using an exogenous ketogenic formula; Behavioral: Online cognitive training
- WaitList Control (Active Comparator): The arm will only use the online cognitive training program Lumosity 3 months after enrollment in the study.
  Interventions: Behavioral: Online cognitive training

INTERVENTIONS:
Behavioral: Modified ketogenic diet using an exogenous ketogenic formula — Participants will follow a modified ketogenic diet consuming a daily exogenous ketogenic meal replacement formula while limiting their carbohydrate intake for 12 weeks.
  Other Names: KetoCal
  Arms: Diet and Cognitive Training
Behavioral: Online cognitive training — Participants will complete a daily session of 5 online cognitive training tasks for 12 weeks.
  Other Names: Lumosity

SUMMARY:
The goal of this clinical trial is to examine feasibility of a cognitive intervention program in blood cancer survivors. The main questions it aims to answer are:

* is it feasible to combine a ketogenic diet supplementation and online cognitive training in an intervention program
* will patients using the combined intervention program have improved cognitive functioning compared to those who don't use it
* how long will the intervention programs effects last

Participants randomized to the intervention arm will consume an exogenous ketogenic supplementation and use an online cognitive training program for 12 weeks, while waitlist arm functions as a control group and will receive the online cognitive training only after a wait period of 12 weeks. Researchers will compare the intervention and waitlist control groups to see if the intervention improves cognitive functioning.

DETAILED DESCRIPTION:
The investigators propose using "off-the-shelf" products in a 12-week multicomponent cognitive intervention program to address the cognitive impairment in outpatient hematologic malignancy survivors. The program includes two components: i) A modified ketogenic diet using an exogenous ketogenic supplementation using the KetoCal product ([https://shop.myketocal.com/product/ketocal-41-lq]) and ii) online cognitive training using Lumosity program (http://www.lumosity.com/).

A ketogenic diet is characterized by high fat, moderate protein and very low carbohydrate intake. Participants will follow a modified ketogenic diet consuming exogenous Ketocal tetrapaks daily to substitute ~700 calories of their daily calorie needs and limit their carbohydrate intake while maintaining an eucaloric diet. The KetoCal is a nutritionally complete, ready-to-feed ketogenic meal replacement product. The study goal is to achieve safe and tolerable levels of mild nutritional ketosis (0.5-2mmol/L betahydroxybutyrate (BHB) blood concentration). Diet education will be provided to participants on how and when to consume the KetoCal formula, foods and beverages consistent with a ketogenic diet and foods and beverages to avoid, and how to measure the ketosis using a breathalyzer daily. Safety and Tolerability monitoring will occur by recording treatment-emergent and/or treatment-related adverse events, regular monitoring of weight and satiety levels, and routine laboratory testing using fasting blood samples at baseline and 12 weeks.

The Lumosity program offers over 60 tasks in game-like format that cover the main cognitive domains: processing speed, working memory, attention and executive function. Training will involve a daily session of 5 training tasks for 12 weeks. Each time the patient is logged in for a session, a customized report will be generated by the Lumosity program to capture performance information.

Participants' cognitive functioning will be assessed at baseline and 12 weeks using objectively measured cognitive function to estimate the preliminary efficacy of intervention program; and at 24 weeks to examine the sustained effects of the multi-component intervention program.

The findings from this project will inform a definitive phase III trial of a multi-component intervention to improve cognitive outcomes in patients with hematologic malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Adult with hematologic malignancy diagnosed at age ≥21 years
* Outpatient at least 3 months from completion of blood or marrow transplant (BMT) or at least 6 months from diagnosis for patients not treated with BMT
* Evidence of mild-to-moderate cognitive impairment using either the Modified Telephone Interview for Mild Cognitive Impairment (TICS-M) or PROMIS 8a short form raw score = 19 -37
* Have daily access to an internet-connected home computer
* Can fluently read and write in English
* Can understand and sign the study-specific Informed Consent Form

Exclusion Criteria:

* History of pre-existing neurological disorder or documented major psychiatric disorder
* Significant auditory, visual, or motor impairments
* History of color blindness
* Participated in neuropsychological intervention within the past 6 months
* Evidence of active chronic graft vs. host disease (GvHD) for allogeneic BMT
* History of pre-existing metabolic disease
* Allergies to soy or milk
* Body Mass Index (BMI) ≤20

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of hematologic malignancy patients completing the 2-arm 12wk randomized wait-listed trial of the multicomponent intervention of modified ketogenic diet and cognitive training | 12 weeks
  Number of participants completing the 12 week intervention
Change in cognitive function global deficit score (GDS) from baseline to 12 wks, comparing patients on the multicomponent active arm to the waitlist arm (prior to receiving cognitive training) | Baseline to 12 weeks
  Change in cognitive function will be measured using the cognitive function global deficit score (GDS) at baseline and 12 weeks comparing both active and waitlist arms. The neuropsychological test battery will include the following tests: D-KEFS Verbal Fluency, DKEFS Color-Word Interference, D-KEFS Trail Making, WAIS-IV Digit-Symbol Coding, WAIS-IV Digit Span, WAIS-IV Letter-Number Sequencing, WMS-IV Logical Memory, CVLT-II). Raw scores from the neuropsychological test battery will be transformed to standardized T-scores (mean=50; SD=10) using published normative data. T-scores will be converted to a deficit score ranging from 0 (no impairment) to 5 (severe impairment) and averaged across all tests to calculate the GDS. A lower GDS score means better cognitive function.

SECONDARY OUTCOMES:
Change in cognitive function global deficit score (GDS) from baseline to 12 wks in patients on the multicomponent active arm compared to change in cognition from 12 wks to 24 wks in patients on the waitlist arm (following receiving cognitive training) | Baseline to 12 weeks for the multicomponent active arm and from 12 weeks to 24 weeks for the waitlist arm
  Change in cognitive function will be measured using cognitive function global deficit score (GDS) at baseline and 12 weeks on the multicomponent active arm and 12 weeks to 24 weeks on the waitlist arm following receiving the cognitive training only. The neuropsychological test battery will include the following tests: D-KEFS Verbal Fluency, DKEFS Color-Word Interference, D-KEFS Trail Making, WAIS-IV Digit-Symbol Coding, WAIS-IV Digit Span, WAIS-IV Letter-Number Sequencing, WMS-IV Logical Memory, CVLT-II). Raw scores from the neuropsychological test battery will be transformed to standardized T-scores (mean=50; SD=10) using published normative data. T-scores will be converted to a deficit score ranging from 0 (no impairment) to 5 (severe impairment) and averaged across all tests to calculate the GDS. A lower GDS score means better cognitive function.
Change in cognitive function global deficit score (GDS) from 12 wks to 24 wks in patients on the multicomponent active arm | 12 weeks to 24 weeks
  Change in cognitive function will be measured using cognitive function global deficit score (GDS) at 12 weeks to 24 weeks on the multicomponent active arm. The neuropsychological test battery will include the following tests: D-KEFS Verbal Fluency, DKEFS Color-Word Interference, D-KEFS Trail Making, WAIS-IV Digit-Symbol Coding, WAIS-IV Digit Span, WAIS-IV Letter-Number Sequencing, WMS-IV Logical Memory, CVLT-II). Raw scores from the neuropsychological test battery will be transformed to standardized T-scores (mean=50; SD=10) using published normative data. T-scores will be converted to a deficit score ranging from 0 (no impairment) to 5 (severe impairment) and averaged across all tests to calculate the GDS. A lower GDS score means better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Sharafeldin, MD, MSc, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States